CLINICAL TRIAL: NCT01798641
Title: Efficacy of Shunt Surgery in Normal Pressure Hydrocephalus: a Randomized Cross-over Study
Brief Title: A Randomized Cross-over Study for Normal Pressure Hydrocephalus
Acronym: ARCS NPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Aesculap, Inc. (Industry); Ohio State University (Other); Rhode Island Hospital (Other); Virginia Commonwealth University (Other); Henry Ford Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NA_00042178
Record Dates: First submitted 2013-01-31; First posted 2013-02-26 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Normal Pressure Hydrocephalus
Keywords: Hydrocephalus; Cross-over
MeSH Terms: conditions — Hydrocephalus, Normal Pressure; Hydrocephalus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Open Shunt (Experimental): The programmable valve, MIETHKE proGAV® / MIETHKE proSA®, will be open at this time. The adjustment is done in the out-patient clinic.
  Interventions: Device: MIETHKE proGAV® / MIETHKE proSA®
- Closed Shunt (Placebo Comparator): The programmable valve, MIETHKE proGAV® / MIETHKE proSA®, will be closed during this time. The adjustment is done in the out-patient clinic.
  Interventions: Device: MIETHKE proGAV® / MIETHKE proSA®

INTERVENTIONS:
Device: MIETHKE proGAV® / MIETHKE proSA® — The programmable shunt will be adjusted through the MIETHKE proGAV® / MIETHKE proSA® valve and crossed over at 6 weeks. The open shunt will be adjusted to be closed. The closed shunt will be adjusted to open.

SUMMARY:
The goal of our study is to verify the effectiveness of the shunt and to identify the most sensitive criteria to select patients for surgery. The study is designed to assess improvement in walking and balance (gait), urinary function and memory after shunting. In addition, the study aims to identify the most accurate and sensitive tools to measure improvement for our patients.

DETAILED DESCRIPTION:
Normal Pressure Hydrocephalus (NPH) causes memory loss, walking, and urinary difficulties. If NPH goes unidentified and untreated it can cause severe disability. The cause of this disease is poorly understood. It may involve damage caused by impaired blood flow in the brain.

The standard methods by which we diagnose patients who have symptoms of NPH are less accurate than desired. Many times patients remain undiagnosed or untreated while others receive treatment due to a false-positive diagnosis.

To treat NPH, a small tube called a 'shunt' can be surgically placed in the brain to drain cerebrospinal fluid (CSF) and help relieve symptoms. Currently, the reported response rates to shunting vary from 31% to 89%. Follow-up studies have shown that the shunts may not work long-term. This could be due to the natural history of the disease, development of other diseases, or due to a short term 'placebo effect' following the shunt placement surgery.

Our group is doing a study of patients with NPH. All participants in this study will have a shunt placed. These shunts are programmable and, once placed, may be opened or closed by the doctor. Programming the shunt does not require an additional surgical procedure. All study participants will be divided into two groups. One group will have their shunts open and draining. The other group will have their shunts closed (not draining). After 6 weeks, the groups will be switched. Those with open shunts will have them closed, and the group with closed, non-draining shunts, will have theirs opened. Participants will not know if their shunts are open (draining) or if they are closed (not draining). Study participants will be followed for two years. Any participants who develop recurrent, new or worsening symptoms will be taken off study and treated according to good medical practice.

The purpose of this study is to (a) look for symptom improvement in response to the draining shunt compared to the non-draining shunt (placebo affect), (b) find 'predictors' that will help doctors identify patients who will respond well to shunt placement, (c) monitor the long-term effects of these shunts, and (d) assess current diagnostic testing to see which methods are most accurate.

Eligibility Criteria:

Inclusion Criteria

1. Age of Patients ( between 60 to 85 years old).
2. Clinically suspected Idiopathic Normal Pressure Hydrocephalus (iNPH) with at least gait impairment.
3. Informed consent from patient.

Exclusion Criteria

1. Etiology for hydrocephalus other than iNPH.
2. Patients not capable of providing an informed consent.
3. History of intra-cerebral hemorrhage.
4. Cardiac Pacemaker.

ELIGIBILITY:
Inclusion Criteria:

* Age of Patients ( between 60 to 85 years old)
* Clinically suspected Normal Pressure Hydrocephalus (NPH) with at least gait impairment
* Informed consent from patient

Exclusion Criteria:

* Etiology for hydrocephalus other than idiopathic normal pressure hydrocephalus
* Patients not capable of providing an informed consent.
* History of intra-cerebral hemorrhage
* Cardiac Pacemaker

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-01; Primary Completion 2017-09-14 (Actual); Study Completion 2017-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Rigamonti, MD FACS, Principal Investigator — Johns Hopkins University; Jennifer Lu, Study Director — Johns Hopkins University
Locations (5):
- United States (5):
  - Johns Hopkins University, Baltimore, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Ohio State University, Columbus, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - Virgina Commonwealth University, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 10 patients (5 from each group) were excluded from the study as further assessment prior to randomization showed significant risk of falls
Groups:
- Open Shunt, Then Closed: The programmable valve, MIETHKE proGAV® / MIETHKE proSA®, will be open at this time. The adjustment is done in the out-patient clinic.
  MIETHKE proGAV® / MIETHKE proSA®: The programmable shunt will be adjusted through the MIETHKE proGAV® / MIETHKE proSA® valve and crossed over at 6 weeks. The open shunt will be adjusted to be closed. The closed shunt will be adjusted to open.
- Closed Shunt, Then Open: The programmable valve, MIETHKE proGAV® / MIETHKE proSA®, will be closed during this time. The adjustment is done in the out-patient clinic.
  MIETHKE proGAV® / MIETHKE proSA®: The programmable shunt will be adjusted through the MIETHKE proGAV® / MIETHKE proSA® valve and crossed over at 6 weeks. The open shunt will be adjusted to be closed. The closed shunt will be adjusted to open.
Period: First Intervention (6 Weeks)
Arm/Group | Open Shunt, Then Closed | Closed Shunt, Then Open
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0
Period: Second Intervention (6 Weeks)
Arm/Group | Open Shunt, Then Closed | Closed Shunt, Then Open
Started | 19 | 19
Completed | 19 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Open Shunt, Then Closed: The programmable valve, MIETHKE proGAV® / MIETHKE proSA®, will be open at this time. The adjustment is done in the out-patient clinic.
  MIETHKE proGAV® / MIETHKE proSA®: The programmable shunt will be adjusted through the MIETHKE proGAV® / MIETHKE proSA® valve and crossed over at 6 weeks. The open shunt will be adjusted to be closed.
- Closed Shunt, Then Open: The programmable valve, MIETHKE proGAV® / MIETHKE proSA®, will be closed during this time. The adjustment is done in the out-patient clinic.
  MIETHKE proGAV® / MIETHKE proSA®: The programmable shunt will be adjusted through the MIETHKE proGAV® / MIETHKE proSA® valve and crossed over at 6 weeks.The closed shunt will be adjusted to open.
- Total: Total of all reporting groups
Arm/Group | Open Shunt, Then Closed | Closed Shunt, Then Open | Total
Number analyzed (Participants) | 19 | 19 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 4 | 6
  >=65 years | 17 | 15 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 11 | 17
  Male | 13 | 8 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 19 | 19 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 19 | 19 | 38
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Tinetti Score on Open Shunt vs. Closed Shunt
Description: The Tinetti tool test measures walking and balance. It is designed to determine an elders risk for falls within the next year. It takes about 8-10 minutes to complete. The patient is asked to complete the gait portion first with the evaluator walking close behind the elder and evaluating gait steppage and drift. The patient is then asked to complete the balance portion with the evaluator again standing close by the patient (towards the right and in front). The patient is then asked to sit and the score is then totaled.The higher the score, the better the performance. Scoring is done on a three point scale with a range on each item of 0-2 with 0 representing the most impairment. Individual scores are then combined to form three scales: a Gait Scale, a Balance Scale and then and overall Gait and Balance score. The maximum score for gait is 12 points while the maximum for Balance is 16 points with a total maximum for the overall score of 28 points.
Time Frame: 6 weeks
Population: Only 10 participants were analyzed from each group. The rest were lost to follow up
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Groups:
- Open Shunt: The programmable valve, MIETHKE proGAV® / MIETHKE proSA®, will be open at this time. The adjustment is done in the out-patient clinic.
  MIETHKE proGAV® / MIETHKE proSA®: The programmable shunt will be adjusted through the MIETHKE proGAV® / MIETHKE proSA® valve and crossed over at 6 weeks. The open shunt will be adjusted to be closed.
- Closed Shunt: The programmable valve, MIETHKE proGAV® / MIETHKE proSA®, will be closed during this time. The adjustment is done in the out-patient clinic.
  MIETHKE proGAV® / MIETHKE proSA®: The programmable shunt will be adjusted through the MIETHKE proGAV® / MIETHKE proSA® valve and crossed over at 6 weeks. The closed shunt will be adjusted to open.
Arm/Group | Open Shunt | Closed Shunt
Number analyzed (Participants) | 10 | 10
score on a scale | 24.50 [23.00 to 27.20] | 26.50 [24.50 to 27.00]

2. Primary Outcome: Timed Up and Go (TUG) Score on Open Shunt vs. Closed Shunt
Description: The TUG evaluation measures walking and balance. The patient is timed while they rise from an arm chair (approximate seat height 46 cm), walk at a comfortable and safe pace to a line on the floor three meters away, turn and walk back to the chair and sit down again. The patient walks through the test once before being timed to become familiar with the test. The subject wears his regular footwear and uses a walking aid (cane or walker) if necessary. A faster time indicates a better functional performance and a score of ≥13.5 seconds is used as a cut-point to identify those at increased risk of falls.
Time Frame: 6 weeks
Population: Only 7 participants were analyzed from the open shunt group. Only 10 were analyzed from the closed shunt group. The rest were lost to follow up
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Open Shunt | Closed Shunt
Number analyzed (Participants) | 7 | 10
seconds | 12.0 [10.00 to 13.70] | 10.5 [8.38 to 15.53]

3. Primary Outcome: Medical College of Virginia (MCV) Gait Grade on Open Shunt vs. Closed Shunt
Description: The MCV gait grade evaluation measures balance and walking. The score ranges from 1 to 6 with higher values suggesting worse gait performance.
Time Frame: 6 weeks
Population: Only 8 from each closed shunt group were analyzed. The rest were lost to follow up
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Closed Shunt: The programmable valve, MIETHKE proGAV® / MIETHKE proSA®, will be closed during this time. The adjustment is done in the out-patient clinic.
  MIETHKE proGAV® / MIETHKE proSA®: The programmable shunt will be adjusted through the MIETHKE proGAV® / MIETHKE proSA® valve and crossed over at 6 weeks.The closed shunt will be adjusted to open.
Arm/Group | Open Shunt | Closed Shunt
Number analyzed (Participants) | 8 | 8
score on a scale | 3.00 [2.00 to 3.00] | 1.50 [1.00 to 3.00]

4. Primary Outcome: Kiefer Score on Open Shunt vs. Closed Shunt
Description: The Kiefer is a modified clinical grading tool that measures the severity of the three key symptoms (mental deficits, gait disturbance, incontinence) and two additional minor symptoms (headache and dizziness). The overall score may reach values between 0 and 24, with higher scores indicating more severe impairment
Time Frame: 6 weeks
Population: Only 11 participants were analyzed from each arm. The remaining were lost to follow up
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Open Shunt | Closed Shunt
Number analyzed (Participants) | 11 | 11
score on a scale | 4 [3 to 6] | 5 [2 to 7]

5. Primary Outcome: Kubo Score on Open Shunt vs. Closed Shunt
Description: The Kubo tool measures your symptoms in three categories: cognitive (attention and memory), gait/balance and urinary function.The score ranges from 0 to 24 with higher scores indicating worse symptoms
Time Frame: 6 weeks
Population: Only 11 participants were analyzed from each group. The rest were lost to follow up.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Open Shunt | Closed Shunt
Number analyzed (Participants) | 11 | 11
score on a scale | 3 [2 to 3] | 4 [2 to 6]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Open Shunt | Closed Shunt
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 4/38 | 0/38
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Shunt (N=38) | Closed Shunt (N=38)
subdural hematoma (Surgical and medical procedures) | 3 (3) | 0 (0)
hygroma (Surgical and medical procedures) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-03-19): https://cdn.clinicaltrials.gov/large-docs/41/NCT01798641/Prot_SAP_000.pdf